CLINICAL TRIAL: NCT06030206
Title: Preparation for Lung Transplant Discussions and Decisions Among People With Cystic Fibrosis
Brief Title: Lung Transplant READY CF 2: A Multi-site RCT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Kathleen Ramos, Associate Professor, School or Medicine, University of Washington
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: STUDY00016585; 1R01NR020470-01A1 (NIH)
Record Dates: First submitted 2023-08-25; First posted 2023-09-08 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Lung Transplantation; Advanced Lung Disease; Decision Support Tool
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Access to an investigator-designed web-based educational resource with information about lung transplant for three months.
  Interventions: Behavioral: Investigator-designed lung transplant education resource (Research Intervention)
- Attention-control (Active Comparator): Access to a publicly available web-based educational resource with information about transplant for three months.
  Interventions: Behavioral: Publicly available transplant education resource (Attention-control)

INTERVENTIONS:
Behavioral: Investigator-designed lung transplant education resource (Research Intervention) — Participants will access the investigator-designed educational resource via their login to a secure website. After three months, participants will gain access to the publicly available website (attention control) and will have an additional three months of access to both of these resources.
  Arms: Intervention
Behavioral: Publicly available transplant education resource (Attention-control) — Participants will access the publicly available education resource via their login to a secure website. After three months, participants will gain access to the investigator-designed educational resource (research intervention) and will have an additional three months of access to both of these resources.
  Arms: Attention-control

SUMMARY:
Lung transplant is an option for treating end-stage lung disease in cystic fibrosis (CF). In the United States, more people with CF and low lung function die each year than undergo lung transplant. More than half of people with CF who die without a lung transplant were never referred for consideration. Patient preference not to undergo lung transplant may account for 25-40% of decisions to defer referral. Rates of death without transplant are higher for people with CF who are members of marginalized communities, including those with Black race, Hispanic ethnicity, or low socioeconomic status. Increasing awareness of lung transplant among people with CF, and promoting understanding of the risks and benefits of transplant, can potentially reduce the number of people with CF who die without a lung transplant.

The CF Foundation (CFF) lung transplant referral guidelines were developed to optimize the timing of referral for lung transplant. These guidelines recommend annual conversations with people with CF once their forced expiratory volume in one second (FEV1) is <50% predicted. Considering lung transplant as a treatment option before it is medically needed will allow more time to learn about lung transplant and address any barriers to lung transplant that may exist.

Investigators are interested in understanding how people with CF use lung transplant educational resources and how one prepares for having discussions and/or making decisions about lung transplant as a treatment option for advanced CF. The purpose of this study is to test whether a research website improves patient preparedness for discussions about lung transplant. Investigators also aim to understand whether there are unique factors that affect people with CF from communities with decreased access to transplant ("communities of concern").

Study involvement will span 6 months and study activities will involve the following:

* Four Zoom research sessions (15-30 minutes each)
* Survey assessments
* Access to a research website that contains educational resources about lung transplant
* Audio recording of a routine CF clinic visit to determine if and how lung transplant is discussed between a participant and his/her/their CF doctor

DETAILED DESCRIPTION:
Lung transplant is an option for treating end-stage lung disease in cystic fibrosis (CF). In the United States, more people with CF with forced expiratory volume in 1 second (FEV1) less than 30% of predicted die each year than undergo lung transplant. More than half of people with CF who die without lung transplant were never referred for consideration, with patients of lower socioeconomic status, Black race, or Hispanic ethnicity disproportionately impacted by limited access to lung transplant. Patient preference not to undergo lung transplant may account for 25-40% of decisions to defer referral. The CF Foundation established lung transplant referral guidelines that recommend people with CF have annual conversations about lung transplant with their CF doctor once their FEV1 is less than 50% of predicted. Considering lung transplant as a treatment option before it is medically needed will allow more time to learn about lung transplant and address any barriers to lung transplant that may exist. By introducing an educational resource that can increase awareness of lung transplant among patients, and promote understanding of the risks and benefits of lung transplant, investigators aim to empower people with CF to take part in shared decision-making with their CF providers, which could reduce the number of people with CF who die without lung transplant.

Based on prior research, investigators developed a novel lung transplant educational resource that addresses patient-identified knowledge gaps and provides personalized educational content to help people with CF prepare for lung transplant discussions and decisions. The web-based educational resource couples real-life CF patient experiences of lung transplant in the form of personal narratives with up-to-date, CF-specific, and guideline-based medical information about lung transplant.

The overall research objectives for this study are to test the efficacy of the investigator-designed educational resource to improve patient preparedness for shared decision making about lung transplant and knowledge about lung transplant, and to evaluate the impact on mental health outcomes (depression and anxiety). The investigator-designed website will be compared to an attention control website to better understand how people with CF use and rank different educational resources' utility. The central hypothesis is that use of the new investigator-designed website that incorporates disease severity data (FEV1 % predicted, supplemental oxygen use, exacerbations) to identify relevant personal narratives and guideline-based educational content will increase a patient's preparedness to engage in discussions about lung transplant beyond the standard information presented on the attention control website.

The study will be a randomized controlled trial. Participants will be randomly assigned 1:1 to one of two educational resources, described above, stratified by FEV1 category (FEV1 30-50% or FEV1 <30% of predicted), CF Center, and whether they are members of the "communities of concern"). The communities of concern include people with Medicaid insurance, high school education or less, Hispanic ethnicity, or Black/Asian/Other race (not White race). Baseline surveys will evaluate knowledge about lung transplant, a Likert scale rating of preparedness for lung transplant discussions, decisional conflict about lung transplant, and mental health. For three months, participants will have access to one of two educational resources via a login to a secure research website. At 2 weeks, there will be a study visit that includes repeated surveys from baseline and the Preparedness for Shared Decision Making (PrepDM) Scale. At 2 to 3 months after randomization, participants will have a routine CF clinic visit, which may be audio-recorded for evaluation of lung transplant discussion. At 3 months after randomization, there will be a study visit that includes repeated surveys from baseline and the PrepDM Scale. After the 3-month study visit, participants will have access to both educational resources via individual login to the secure research website. At 6-months, there will be a study visit to repeat the surveys. Throughout the 6-months and for a long-term follow up period of 4 years, web analytics will be captured at the individual level to determine usage patterns for both educational resources.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cystic fibrosis
* FEV1 less than 50% of predicted

Exclusion Criteria:

* People who are unable to provide informed consent
* People who are lung transplant recipients
* Unable to read or understand English or Spanish to complete surveys or access the website (currently only available in English and Spanish)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2023-09-06 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Preparedness for Shared Decision Making (PrepDM) Scale | Measured at the 3-month study visit
  The primary endpoint is an intention-to-treat assessment of the difference in mean Preparedness for Shared Decision Making (PrepDM) Scale in the intervention versus attention-control arms of the study at the 3-month study visit using linear mixed models. Scores range on a scale from 0 to 100 with higher scores indicating a higher perceived level of preparation for decision making.

SECONDARY OUTCOMES:
Confidence-weighted true false knowledge about lung transplant (14-question investigator-designed survey) | Measured at 3-month study visit
  Difference in mean change in confidence-weighted true false (CTF) knowledge score will be measured in the intervention versus control arms of the study using linear mixed models. CTF scoring adds points for certainty in correct responses and deducts points for certainty in incorrect responses. Participants receive +2 points when "sure" about a correct response, +1 if unsure about a correct response, -1 if unsure about an incorrect response and -2 if sure about an incorrect response. For a 14-item knowledge test, the maximum score is +28 and the minimum score is -28, with higher scores indicating more knowledge about lung transplant.
Decisional Conflict Scale | Baseline to 3-month study visit
  Decisional Conflict Scale change will be measured from the baseline study visit to the 3-month study visit. The intention-to-treat analysis will compare mean change in the Decisional Conflict Scale between the intervention and control arms of the study. Scores range from 0 [no decisional conflict] to 100 [extremely high decisional conflict].
Likert-scale rating of preparedness to discuss lung transplant (0-4) | Measured at 3-month study visit
  Likert rating of preparedness to discuss lung transplant will be measured at each study visit (0=Don't know, 1= Not at all prepared, 2 = A little prepared, 3 = Moderately prepared, 4 = Very prepared). The intention-to-treat analysis will compare mean change in Likert-scale rating between the intervention and attention-control arms of the study using linear mixed models.
Patient Health Questionnaire (PHQ-9) | Measured at 3-month study visit
  PHQ-9 is a scale that measures symptoms of depression in the prior 2 weeks on a 0-27 scale, with higher scores indicating worsening depression and a score of 10 or higher consistent with a diagnosis of depression. The intention-to-treat analysis will compare mean change in PHQ-9 between the intervention and attention-control arms of the study using linear mixed models. Investigators will also determine the proportion with new PHQ-9 score greater than or equal to 10 in each arm.
Generalized Anxiety Disorder 7-item (GAD-7) Scale | Measured at 3-month study visit
  GAD-7 is a scale that measures symptoms of anxiety in the prior 2 weeks on a 0-21 scale, with higher scores indicating worsening anxiety and a score of 10 or higher consistent with a diagnosis of generalized anxiety disorder. The intention-to-treat analysis will compare mean change in GAD-7 between the intervention and attention-control arms of the study using linear mixed models. Investigators will also determine the proportion with new GAD-7 score greater than or equal to 10 in each arm.

OTHER OUTCOMES:
6-month assessment of Preparedness for Shared Decision Making (PrepDM) Scale | Measured at 6-month study visit
  The PrepDM Scale will be measured for all participants with respect to the investigator-designed educational resource (research intervention) and mean score will be compared for participants in the intervention (6 months of exposure) versus control arms (3 months of exposure) using linear mixed models. PrepDM scores range on a scale from 0 to 100 with higher scores indicating a higher perceived level of preparation for decision making.
6-month assessment for confidence-weighted true false knowledge about lung transplant (14-question investigator-designed survey) | Measured at 6-month study visit
  Change in confidence-weighted true false knowledge about lung transplant (14-question investigator-designed survey) will be assessed from baseline to 6-months and from 3-month to 6-month study visits. Mean difference in the change in knowledge score will be compared between study arms for the two time periods (0 to 6 months and 3 to 6 months). Higher scores indicate more knowledge about lung transplant.
6-month assessment for Decisional Conflict Scale | Measured at 6-months study visit
  Change in Decisional Conflict Scale will be assessed from baseline to 6-months and from 3-month to 6-month study visits. Mean difference in the change in Decisional Conflict Scale will be compared between study arms for the two time periods (0 to 6 months and 3 to 6 months). Scores range from 0 [no decisional conflict] to 100 [extremely high decisional conflict].
6-month assessment for Likert-scale rating of preparedness to discuss lung transplant | Measured at baseline, 3-month and 6-month study visits
  Evaluate the proportion "Very prepared" at baseline, 3-months and 6-months in the intervention and control arms. Compare proportions across study arms at each time point.
Time spent using the research website | Baseline to 3-month study visit
  Average time spent using the research website from baseline to 3-months will be compared across study arms. Further, time spent using the investigator-designed website will be assessed as a predictor of: 1. change in confidence-weighted true false knowledge about lung transplant (14-question investigator-designed survey) from baseline to 3-month study visit, 2. change in Likert preparedness from baseline to 3-month study visit, 3. change in Decisional Conflict Scale from baseline to 3-month study visit, and 4. mean PrepDM Scale at 3-months.
Between-arm comparisons of Shared Decision Making Questionnaire (SDM-Q-9) | Routine CF Clinic visit during the trial
  The analysis will be an intention-to-treat assessment of the difference in mean Shared Decision Making Questionnaire (SDM-Q-9) in the intervention versus attention-control arms of the study at the routine CF Clinic visit using linear mixed models. The SDM-Q-9 scale has a range of (0 to 45), with higher scores indicating higher quality of shared decision making from the patient's perspective. A change in SDM-Q-9 of 12 to 15 has been considered clinically meaningful.
Between-arm comparisons of Shared Decision Making Questionnaire for physicians (SDM-Q-doc) | Routine CF Clinic visit during the trial
  The analysis will be an intention-to-treat assessment of the difference in mean Shared Decision Making Questionnaire for physicians (SDM-Q-doc) in the intervention versus attention-control arms of the study at the routine CF Clinic visit using linear mixed models. The SDM-Q-doc scale has a range of (0 to 45), with higher scores indicating higher quality of shared decision making from the physician's perspective.
Preparedness for Shared Decision Making (PrepDM) Scale among members of communities of concern. | Measured at 3-month study visit
  In a prespecified subgroup analysis, investigators will assess the Preparedness for Shared Decision Making (PrepDM) Scale at 3 months within the cohort of participants who are members of communities of concern. This is an intention-to-treat assessment of the difference in mean Preparedness for Shared Decision Making (PrepDM) Scale in the intervention versus attention-control arms of the study at the 3-month study visit using linear mixed models in the subset of individuals who are members of communities of concern (Medicaid insurance, high-school education or less, Hispanic ethnicity, Black/Asian/Other race). Scores range on a scale from 0 to 100 with higher scores indicating a higher perceived level of preparation for decision making.
Decisional Conflict Scale among members of communities of concern. | Baseline to 3-month study visit
  In a prespecified subgroup analysis, investigators will assess Decisional Conflict Scale change within the cohort of participants who are members of communities of concern (Medicaid insurance, high-school education or less, Hispanic ethnicity, Black/Asian/Other race). Decisional Conflict Scale change will be measured from the baseline study visit to the 3-month study visit. The intention-to-treat analysis will compare mean change in the Decisional Conflict Scale between the intervention and control arms of the study in the subset of individuals who are members of communities of concern. Scores range from 0 [no decisional conflict] to 100 [extremely high decisional conflict].
Confidence-weighted true false knowledge about lung transplant (14-question investigator-designed survey) among members of communities of concern. | Baseline to 3-month study visit
  In a prespecified subgroup analysis, investigators will assess the difference in mean change from baseline to 3 months in Confidence-weighted true false (CTF) knowledge score will be measured in the intervention versus control arms of the study using linear mixed models within the cohort of participants who are members of communities of concern (Medicaid insurance, high-school education or less, Hispanic ethnicity, Black/Asian/Other race). CTF scoring adds points for certainty in correct responses and deducts points for certainty in incorrect responses. Participants receive +2 points when "sure" about a correct response, +1 if unsure about a correct response, -1 if unsure about an incorrect response and -2 if sure about an incorrect response. For a 14-item knowledge test, the maximum score is +28 and the minimum score is -28, with higher scores indicating more knowledge about lung transplant.
Likert rating of preparedness to discuss lung transplant among members of communities of concern. | Baseline to 3-month study visit
  In a prespecified subgroup analysis, investigators will assess change from baseline to 3 months in Likert rating of preparedness to discuss lung transplant within the cohort of participants who are members of communities of concern (Medicaid insurance, high-school education or less, Hispanic ethnicity, Black/Asian/Other race). The intention-to-treat analysis will compare mean change in the Likert rating of preparedness to discuss lung transplant between the intervention and control arms of the study in the subset of individuals who are members of communities of concern. Likert rating of preparedness to discuss lung transplant will be measured at each study visit (0=Don't know, 1= Not at all prepared, 2 = A little prepared, 3 = Moderately prepared, 4 = Very prepared).
Evaluation of CF Clinic audio-recordings and transcripts | Routine CF Clinic visit (at least 6 weeks after randomization/until 3-Month Session) during the trial
  Recordings will be listened to by at least two members of the study team for assessment or implicit bias (e.g. speech rate, verbal dominance) and whether the topic of LTx is raised with different frequency among participants from communities of concern.

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Ramos, MD, MSc, Principal Investigator — University of Washington
Locations (11):
- United States (11):
  - University of California at Los Angeles (UCLA), Los Angeles, California
  - National Jewish Health, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - University of Kansas, Kansas City, Kansas
  - Maine Health, Portland, Maine
  - Johns Hopkins University, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - University of Cincinnati, Cincinnati, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - University of Washington Medical Center - Montlake, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) may be shared with other researchers for secondary analyses with the approval of the appropriate Human Subjects Division(s) and the study's principal investigator (PI).
Supporting Information: Study Protocol, ICF
Time Frame: Data will become available after publication of the results of the primary analyses of the study. The data will be available for up to 3 years after the end of the study.
Access Criteria: Qualified researchers with appropriate clinical research training and/or mentorship will be allowed to have access to IPD after approval is obtained from Human Subjects Division(s) and the study PI.

REFERENCES:
- [Background] Ramos KJ, Smith PJ, McKone EF, Pilewski JM, Lucy A, Hempstead SE, Tallarico E, Faro A, Rosenbluth DB, Gray AL, Dunitz JM; CF Lung Transplant Referral Guidelines Committee. Lung transplant referral for individuals with cystic fibrosis: Cystic Fibrosis Foundation consensus guidelines. J Cyst Fibros. 2019 May;18(3):321-333. doi: 10.1016/j.jcf.2019.03.002. Epub 2019 Mar 27. PMID 30926322
- [Background] Hartzler AL, Bartlett LE, Hobler MR, Reid N, Pryor JB, Kapnadak SG, Berry DL, Lober WB, Goss CH, Ramos KJ; Take on Transplant Study Group. Take on transplant: human-centered design of a patient education tool to facilitate informed discussions about lung transplant among people with cystic fibrosis. J Am Med Inform Assoc. 2022 Dec 13;30(1):26-37. doi: 10.1093/jamia/ocac176. PMID 36173364

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-09): https://cdn.clinicaltrials.gov/large-docs/06/NCT06030206/Prot_SAP_000.pdf
  • Informed Consent Form (2023-08-29): https://cdn.clinicaltrials.gov/large-docs/06/NCT06030206/ICF_001.pdf